CLINICAL TRIAL: NCT02407756
Title: A Phase 2a Study Investigating the Safety, Pharmacokinetics, Immunogenicity, and Exploratory Efficacy of Dupilumab in Patients Aged ≥6 to <18 Years With Atopic Dermatitis
Brief Title: A Study to Determine the Safety and Tolerability of Dupilumab (REGN668/SAR231893) in Patients Aged ≥6 to <18 Years With Atopic Dermatitis (Eczema)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R668-AD-1412
Record Dates: First submitted 2015-03-31; First posted 2015-04-03 (Estimated); Results first posted 2020-10-05 (Actual); Last update posted 2020-11-27 (Actual); Status verified 2020-11

CONDITIONS: Atopic Dermatitis
Keywords: Eczema
MeSH Terms: conditions — Dermatitis, Atopic; Eczema | interventions — dupilumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cohort 1 (Experimental): Cohort 1 will receive dupilumab dosing regimen 1
  Interventions: Drug: Dupilumab
- Cohort 2 (Experimental): Cohort 2 will receive dupilumab dosing regimen 2
  Interventions: Drug: Dupilumab

INTERVENTIONS:
Drug: Dupilumab
  Other Names: REGN668(SAR231893)

SUMMARY:
The primary objective of the study is to characterize the safety and pharmacokinetics (PK) of dupilumab in pediatric patients with moderate-to-severe atopic dermatitis (AD) (for adolescents ≥12 to <18 years of age) or severe AD (for children ≥6 to <12 years of age).

The secondary objective of the study is to explore the immunogenicity and efficacy of dupilumab in pediatric patients with moderate-to-severe AD (for adolescents ≥12 to <18 years of age) or severe AD (for children ≥6 to <12 years of age).

ELIGIBILITY:
Key Inclusion Criteria:

1. Male or female patients ≥6 to <18 years of age with a diagnosis of 1. Atopic Dermatitis whose disease cannot be adequately controlled with topical medications
2. Minimum disease severity, as defined by Investigator's Global Assessment (IGA)

   1. IGA = 3 or 4 in adolescents ≥12 to <18 year of age
   2. IGA = 4 in children ≥6 to <12 years of age

Key Exclusion Criteria:

1. Recent treatment (within specific time windows before the baseline visit) with systemic immunosuppressive agents for eg. Systemic corticosteroids, live (attenuated) vaccines and other investigational drugs including biologics
2. History of any of the following infections:

   1. Any systemic infection requiring treatment within 4 weeks before the baseline visit
   2. Superficial skin infections within 1 week before the baseline visit
   3. Known history of HIV infection
   4. History of seropositivity to hepatitis B or C screening tests
   5. History of clinical endoparasitosis (ie, helminthic infection) within 12 months before the baseline visit, or high risk of helminthic infection, unless subsequent medical assessments (e.g. stool exam, blood tests, etc.) have ruled out the possibility of parasite infection/infestation
3. History of malignancy within 5 years before the baseline visit
4. Persistent (confirmed by repeated tests ≥2 weeks apart) elevated transaminases (alanine aminotransferase [ALT] and/or aspartate aminotransferase [AST]) more than 3 times the upper limit of normal (ULN) during the screening period
5. Presence of any severe concomitant illness(es) that, in the investigator's judgment, would adversely affect the patient's participation in the study
6. Presence of skin comorbidities that may interfere with study assessments
7. Females patients who are pregnant or breastfeeding
8. Female patients who are of reproductive potential and are sexually active, who are unwilling to use adequate methods of contraception

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 78 (Actual)
Dates: Start 2015-03-31 (Actual); Primary Completion 2016-03-31 (Actual); Study Completion 2016-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (26):
- Canada (4):
  - Markham, Ontario
  - Peterborough, Ontario
  - Waterloo, Ontario
  - Windsor, Ontario
- Czechia (2):
  - Kutná Hora
  - Prague
- Germany (9):
  - Dresden
  - Frankfurt
  - Gera
  - Hamburg
  - Kiel
  - Lübeck
  - Munich
  - Münster
  - Tübingen
- Hungary (4):
  - Kaposvár
  - Miskolc
  - Szeged
  - Szolnok
- Poland (5):
  - Katowice
  - Krakow
  - Lodz
  - Warsaw
  - Wroclaw
- United Kingdom (2):
  - Manchester
  - Sheffield

REFERENCES:
- [Derived] Blauvelt A, Guttman-Yassky E, Paller AS, Simpson EL, Cork MJ, Weisman J, Browning J, Soong W, Sun X, Chen Z, Kosloski MP, Kamal MA, Delevry D, Chuang CC, O'Malley JT, Bansal A. Long-Term Efficacy and Safety of Dupilumab in Adolescents with Moderate-to-Severe Atopic Dermatitis: Results Through Week 52 from a Phase III Open-Label Extension Trial (LIBERTY AD PED-OLE). Am J Clin Dermatol. 2022 May;23(3):365-383. doi: 10.1007/s40257-022-00683-2. Epub 2022 May 14. PMID 35567671
- [Derived] Cork MJ, Thaci D, Eichenfield LF, Arkwright PD, Hultsch T, Davis JD, Zhang Y, Zhu X, Chen Z, Li M, Ardeleanu M, Teper A, Akinlade B, Gadkari A, Eckert L, Kamal MA, Ruddy M, Graham NMH, Pirozzi G, Stahl N, DiCioccio AT, Bansal A. Dupilumab in adolescents with uncontrolled moderate-to-severe atopic dermatitis: results from a phase IIa open-label trial and subsequent phase III open-label extension. Br J Dermatol. 2020 Jan;182(1):85-96. doi: 10.1111/bjd.18476. Epub 2019 Oct 8. PMID 31595499

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 25 sites in 6 countries. A total of 88 participants were screened, and of those, 78 participants were randomized with 77 being treated. Ten participants were screen failures as 5 were due to exclusion criteria met & inclusion criteria not met, 4 participants withdrew consent and 1 participant was lost to follow-up.
Pre-assignment Details: A total of 40 adolescents (aged ≥12 to <18 years) and 38 children (aged ≥6 to <12 years) were enrolled and randomized to 2 sequential ascending dose cohorts: Cohort 1 (2 mg/kg) and Cohort 2 (4 mg/kg).
Groups:
- Dupilumab 2mg/kg: Adolescents: Dupilumab 2 mg/kg as a single dose on Day 1 followed by 8-week PK sampling period then 4 repeated doses weekly in subjects aged between ≥12 to <18 years.
- Dupilumab 2mg/kg: Children: Dupilumab 2 mg/kg as a single dose on Day 1 followed by 8-week PK sampling period then 4 repeated doses weekly in subjects aged between ≥6 to <12 years.
- Dupilumab 4mg/kg: Adolescents: Dupilumab 4 mg/kg as a single dose on Day 1 followed by 8-week PK sampling period then 4 repeated doses weekly in subjects aged between ≥12 to <18 years.
- Dupilumab 4mg/kg: Children: Dupilumab 4 mg/kg as a single dose on Day 1 followed by 8-week PK sampling period then 4 repeated doses weekly in subjects aged between ≥6 to <12 years.
Period: Overall Study
Arm/Group | Dupilumab 2mg/kg: Adolescents | Dupilumab 2mg/kg: Children | Dupilumab 4mg/kg: Adolescents | Dupilumab 4mg/kg: Children
Started | 20 | 18 | 20 | 19
Treated | 20 | 18 | 20 | 19
Completed | 20 | 18 | 20 | 19
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dupilumab 2mg/kg: Adolescents | Dupilumab 2mg/kg: Children | Dupilumab 4mg/kg: Adolescents | Dupilumab 4mg/kg: Children | Total
Number analyzed (Participants) | 20 | 18 | 20 | 19 | 77
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.7 (2.01) | 8.2 (1.62) | 14.3 (1.66) | 8.2 (1.99) | 11.5 (3.64)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 9 | 11 | 8 | 39
  Male | 9 | 9 | 9 | 11 | 38
Ethnicity [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 1 | 1
  Not Hispanic or Latino | 20 | 18 | 20 | 18 | 76
Race [Count of Participants; unit: Participants]
  White | 17 | 17 | 15 | 18 | 67
  Black or African American | 0 | 0 | 1 | 1 | 2
  Asian | 2 | 0 | 3 | 0 | 5
  Other | 1 | 1 | 1 | 0 | 3
Number of Subjects with Investigator Global Assessment (IGA) score of 3 or 4 [Count of Participants; unit: Participants] — IGA is an assessment scale used to determine severity of AD and clinical response to treatment on a 5-point scale (0 = clear; 1 = almost clear; 2 = mild; 3 = moderate; 4 = severe) based on erythema and papulation/ infiltration. Therapeutic response is an IGA score of 0 (clear) or 1 (almost clear). Analysis was performed on SAF.
  Participants
    IGA score of 3 | 8 | 1 | 11 | 0 | 20
    IGA score of 4 | 12 | 17 | 9 | 19 | 57
Eczema Area and Severity Index (EASI) score [Mean (Standard Deviation); unit: Score on a scale] — The EASI score was used to measure the severity and extent of atopic dermatitis (AD) and measures erythema, infiltration, excoriation and lichenification on 4 anatomic regions of the body: head, trunk, upper and lower extremities. The total EASI score ranges from 0 to 72 points, with the higher scores reflecting the worse severity of AD. Analysis was performed on Safety Analysis set (SAF).
  Score on a scale | 34.8 (17) | 32.9 (15.53) | 28.6 (14.7) | 38.8 (18.64) | 33.7 (16.62)
Pruritus Numerical Rating Scale (NRS) [Mean (Standard Deviation); unit: Score on a scale] — Pruritus NRS scale is an assessment tool that is used to report the intensity of subject's pruritus (itch), both maximum and average intensity, during a 24-hour recall period. Subjects were asked the following question: how would a subject rate his itch at the worst moment during the previous 24 hours (for maximum itch intensity on a scale of 0 - 10 [0 = no itch; 10 = worst itch imaginable]). Weekly average obtained in the 7-day period prior to the baseline visit. Analysis was performed on SAF.
  Score on a scale | 6.1 (2.47) | 6.4 (2.23) | 6.9 (2.21) | 6.7 (2.35) | 6.5 (2.29)
Body Surface Area (BSA) Involvement with Atopic Dermatitis (AD) [Mean (Standard Deviation); unit: Percentage of body surface area] — BSA affected by AD was assessed for each section of the body (the possible highest score for each region was: head and neck [9%], anterior trunk [18%], back [18%], upper limbs [18%], lower limbs [36%], and genitals [1%]). It was reported as a percentage of all major body sections combined. Analysis was performed on SAF.
  Percentage of body surface area | 52.2 (24.78) | 59 (22.49) | 45.9 (25.34) | 62.3 (30.34) | 54.6 (26.19)
SCORing Atopic Dermatitis (SCORAD) Score [Mean (Standard Deviation); unit: Score on a scale] — SCORAD is a clinical tool for assessing the severity of atopic dermatitis developed by the European Task Force on Atopic Dermatitis ("Severity scoring of atopic dermatitis: the SCORAD index. Consensus Report of the European Task Force on Atopic Dermatitis". Dermatology (Basel) 186 (1): 23-31. 1993). Extent and intensity of eczema as well as subjective signs (insomnia, etc.) are assessed and scored. Total score ranges from 0 [absent disease] to 103 [severe disease]). Analysis was performed on SAF.
  Score on a scale | 68 (13.19) | 66.4 (13.06) | 63 (14.43) | 72.7 (12.96) | 67.5 (13.64)

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics (PK) of Dupilumab: Maximum Plasma Concentration Observed (Cmax) After Single Administration
Description: Peak dupilumab concentration in serum following single dose administration. Analysis was performed on PK analysis set that included all treated subjects who received the study medication and had at least 1 quantified (non-missing) result for dupilumab concentration following the first dose of the study drug.
Time Frame: Day 2, 4, 8, 15, 22, 29, 36, 43, and 50
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Dupilumab 2mg/kg: Adolescents | Dupilumab 2mg/kg: Children | Dupilumab 4mg/kg: Adolescents | Dupilumab 4mg/kg: Children
Number analyzed (Participants) | 20 | 18 | 20 | 19
mg/L | 9.91 (2.15) [lower limit 2.15] | 14.3 (5.9) [lower limit 5.9] | 23.1 (8.71) [lower limit 8.71] | 32.4 (7.04) [lower limit 7.04]

2. Primary Outcome: PK of Dupilumab: Area Under the Plasma Concentration Versus Time Curve (AUClast) After Single Administration
Description: Mean AUC estimates were calculated using mean concentration data at each time point, using a non-compartmental approach (NCA). Calculated AUClast (computed from time zero to the time of the last positive concentration) are presented. Analysis was performed on PK analysis set that included all treated subjects who received the study medication and had at least 1 quantified (non-missing) result for dupilumab concentration following the first dose of the study drug.
Time Frame: Day 2, 4, 8, 15, 22, 29, 36, 43, and 50
Measure: Mean (Standard Deviation); unit: Day*mg/L
Arm/Group | Dupilumab 2mg/kg: Adolescents | Dupilumab 2mg/kg: Children | Dupilumab 4mg/kg: Adolescents | Dupilumab 4mg/kg: Children
Number analyzed (Participants) | 20 | 18 | 20 | 19
Day*mg/L | 104 (NA) — Standard deviation is not available, as AUC was not calculated individually due to the sparse nature of the data collected per participant, rendering individual estimates inaccurate | 160 (NA) — Standard deviation is not available, as AUC was not calculated individually due to the sparse nature of the data collected per participant, rendering individual estimates inaccurate | 362 (NA) — Standard deviation is not available, as AUC was not calculated individually due to the sparse nature of the data collected per participant, rendering individual estimates inaccurate | 330 (NA) — Standard deviation is not available, as AUC was not calculated individually due to the sparse nature of the data collected per participant, rendering individual estimates inaccurate

3. Primary Outcome: PK of Dupilumab: Trough Dupilumab Concentration in Serum (Ctrough) Before 3rd and 4th Repeated Dose
Description: Analysis was performed on PK analysis set that included all treated subjects who received the study medication and had at least 1 quantified (non-missing) result for dupilumab concentration following the first dose of study drug.
Time Frame: Pre-dose on Day 71 and Day 85
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Dupilumab 2mg/kg: Adolescents | Dupilumab 2mg/kg: Children | Dupilumab 4mg/kg: Adolescents | Dupilumab 4mg/kg: Children
Number analyzed (Participants) | 20 | 18 | 20 | 19
mg/L
  Day 71 | 10.4 (7.16) | 17.2 (8.44) | 32.8 (18.9) | 42.1 (19.4)
  Day 85 | 18.5 (12.4) | 28 (12.9) | 58.8 (24.4) | 60.3 (36.3)

4. Secondary Outcome: Percent Reduction From Baseline in Eczema Area and Severity Index (EASI) at Week 12
Description: The EASI score was used to measure the severity and extent of atopic dermatitis (AD) and measures erythema, infiltration, excoriation and lichenification on 4 anatomic regions of the body: head, trunk, upper and lower extremities. The total EASI score ranges from 0 to 72 points, with the higher scores reflecting the worse severity of AD. Analysis was performed on safety analysis set (SAF) that included all subjects who received any study drug. Data after rescue treatment use during the Part B period were set to missing, then missing values were imputed by last observation carried forward (LOCF).
Time Frame: Baseline to Week 12 (one week after last dose)
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Dupilumab 2mg/kg: Adolescents | Dupilumab 2mg/kg: Children | Dupilumab 4mg/kg: Adolescents | Dupilumab 4mg/kg: Children
Number analyzed (Participants) | 20 | 18 | 20 | 19
percent change | -66.4 (29.25) [lower limit 29.25] | -76.2 (25.48) [lower limit 25.48] | -69.7 (24.48) [lower limit 24.48] | -63.4 (25.37) [lower limit 25.37]

5. Secondary Outcome: Percent Reduction From Baseline in SCORing Atopic Dermatitis (SCORAD) Score at Week 12
Description: SCORAD is a clinical tool for assessing the severity of atopic dermatitis developed by the European Task Force on Atopic Dermatitis ("Severity scoring of atopic dermatitis: the SCORAD index. Consensus Report of the European Task Force on Atopic Dermatitis". Dermatology (Basel) 186 (1): 23-31. 1993). Extent and intensity of eczema as well as subjective signs (insomnia, etc.) are assessed and scored. Total score ranges from 0 [absent disease] to 103 [severe disease]). Analysis was performed on SAF. Data after rescue treatment use during the Part B period were set to missing, then missing values were imputed by LOCF.
Time Frame: Baseline to Week 12 (one week after last dose)
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Dupilumab 2mg/kg: Adolescents | Dupilumab 2mg/kg: Children | Dupilumab 4mg/kg: Adolescents | Dupilumab 4mg/kg: Children
Number analyzed (Participants) | 20 | 18 | 20 | 19
percent change | -47.7 (27.27) [lower limit 27.27] | -57.5 (23.1) [lower limit 23.1] | -43.4 (25.38) [lower limit 25.38] | -46.9 (24.31) [lower limit 24.31]

6. Secondary Outcome: Percent Reduction From Baseline in Pruritus Numerical Rating Scale (NRS) at Week 12
Description: Pruritus NRS scale is an assessment tool that is used to report the intensity of subject's pruritus (itch), both maximum and average intensity, during a 24-hour recall period. Subjects were asked the following question: how would a subject rate his itch at the worst moment during the previous 24 hours (for maximum itch intensity on a scale of 0 - 10 [0 = no itch; 10 = worst itch imaginable]). Analysis was performed on SAF. Data after rescue treatment use during the Part B period were set to missing, then missing values were imputed by LOCF.
Time Frame: Baseline to Week 12 (one week after last dose)
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Dupilumab 2mg/kg: Adolescents | Dupilumab 2mg/kg: Children | Dupilumab 4mg/kg: Adolescents | Dupilumab 4mg/kg: Children
Number analyzed (Participants) | 20 | 18 | 20 | 19
Percent change | -30.8 (68.35) [lower limit 68.35] | -41.6 (35.32) [lower limit 35.32] | -37.6 (34.42) [lower limit 34.42] | -39.6 (40.88) [lower limit 40.88]

7. Secondary Outcome: Percentage of Subjects With Investigator Global Assessment (IGA) Score of "0" or "1" (Clear or Almost Clear) at Week 12
Description: IGA is an assessment scale used to determine severity of AD and clinical response to treatment on a 5-point scale (0 = clear; 1 = almost clear; 2 = mild; 3 = moderate; 4 = severe) based on erythema and papulation/infiltration. Therapeutic response is an IGA score of 0 (clear) or 1 (almost clear). Analysis was performed on SAF. Subjects with rescue treatment usage during the Part B period were specified as non-responders from the time the rescue was used.
Time Frame: Week 12
Measure: Number; unit: Percentage of subjects
Arm/Group | Dupilumab 2mg/kg: Adolescents | Dupilumab 2mg/kg: Children | Dupilumab 4mg/kg: Adolescents | Dupilumab 4mg/kg: Children
Number analyzed (Participants) | 20 | 18 | 20 | 19
Percentage of subjects | 10 | 16.7 | 35 | 21.1

8. Secondary Outcome: Percent Reduction From Baseline in Body Surface Area (BSA) at Week 12
Description: Body surface area affected by AD was assessed for each section of the body (the possible highest score for each region was: head and neck [9%], anterior trunk [18%], back [18%], upper limbs [18%], lower limbs [36%], and genitals [1%]). It was reported as a percentage of all major body sections combined. Analysis was performed on SAF.
Time Frame: Baseline to Week 12
Population: Here "Number of participants analyzed" = number of participants who were evaluated for this specific outcome measure.
Measure: Mean (Standard Deviation); unit: Percentage of body surface area
Arm/Group | Dupilumab 2mg/kg: Adolescents | Dupilumab 2mg/kg: Children | Dupilumab 4mg/kg: Adolescents | Dupilumab 4mg/kg: Children
Number analyzed (Participants) | 19 | 16 | 19 | 19
Percentage of body surface area | -61 (31.08) [lower limit 31.08] | -70 (31.93) [lower limit 31.93] | -60.4 (34.04) [lower limit 34.04] | -50 (30.8) [lower limit 30.8]

ADVERSE EVENTS:
Time Frame: All Adverse Events (AEs) were collected from signature of the informed consent form up to the final visit (Week 20) regardless of seriousness or relationship to investigational product.
Description: Treatment Emergent Adverse Events (TEAEs) that developed/ worsened during the treatment and follow-up period (time period from the administration of first dose of study drug to End of Study (EOS) visit [8 weeks after the last dose). Analysis was performed on SAF.
Groups:
- Dupilumab 2mg/kg: Adolescents: Dupilumab 2 mg/kg as a single dose on Day 1 followed by 8-week PK sampling period, then 4 repeated doses weekly in subjects aged between ≥12 to <18 years.
- Dupilumab 2mg/kg: Children: Dupilumab 2 mg/kg as a single dose on Day 1 followed by 8-week PK sampling period, then 4 repeated doses weekly in subjects aged between ≥6 to <12 years.
- Dupilumab 4 mg/kg: Adolescents: Dupilumab 4 mg/kg as a single dose on Day 1 followed by 8-week PK sampling period, then 4 repeated doses weekly in subjects aged between ≥12 to <18 years.
- Dupilumab 4 mg/kg: Children: Dupilumab 4 mg/kg as a single dose on Day 1 followed by 8-week PK sampling period), then 4 repeated doses weekly in subjects aged between ≥6 to <12 years.
Arm/Group | Dupilumab 2mg/kg: Adolescents | Dupilumab 2mg/kg: Children | Dupilumab 4 mg/kg: Adolescents | Dupilumab 4 mg/kg: Children
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/18 | 0/20 | 0/19
Serious Adverse Events (participants affected / at risk) | 1/20 | 0/18 | 1/20 | 2/19
Other Adverse Events (participants affected / at risk) | 11/20 | 11/18 | 16/20 | 18/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dupilumab 2mg/kg: Adolescents (N=20) | Dupilumab 2mg/kg: Children (N=18) | Dupilumab 4 mg/kg: Adolescents (N=20) | Dupilumab 4 mg/kg: Children (N=19)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Staphylococcal skin infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthritis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dermatitis infected (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dupilumab 2mg/kg: Adolescents (N=20) | Dupilumab 2mg/kg: Children (N=18) | Dupilumab 4 mg/kg: Adolescents (N=20) | Dupilumab 4 mg/kg: Children (N=19)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Cyanosis (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eosinophilia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Conjunctivitis allergic (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Dermoid cyst (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aphthous stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cheilitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 3 (3)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Chills (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Pyrexia (General disorders) | 2 (4) | 0 (0) | 0 (0) | 2 (2)
Injection site urticaria (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Injection site swelling (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Injection site irritation (General disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Injection site erythema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Feeling of body temperature change (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Food allergy (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bacterial disease carrier (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Allergic oedema (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Croup infectious (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dermatitis infected (Infections and infestations) | 0 (0) | 1 (1) | 2 (4) | 2 (5)
Ear infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Folliculitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gingivitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Herpes simplex (Infections and infestations) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Molluscum contagiosum (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Laryngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Herpes virus infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 2 (3) | 5 (9) | 8 (11) | 10 (11)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhinitis (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 2 (2)
Pharyngitis bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pharyngitis streptococcal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Paronychia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin bacterial infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Skin candida (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 1 (1) | 1 (1) | 1 (1)
Tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Animal bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bone contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Post procedural inflammation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Increased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Protein urine present (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Epiphysiolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Akathisia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (2) | 1 (1) | 1 (1) | 2 (3)
Lethargy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Depressed mood (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 1 (2) | 7 (8)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (2)
Nasal disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alopecia areata (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 2 (2) | 5 (11) | 3 (6) | 5 (10)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin erosion (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain of skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Solar dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vitiligo (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator has the right to independently publish study results from the investigator's site after a multi-center publication, or a defined period after the completion of the study by all sites. The investigator must provide the sponsor a copy of any such publication derived from the study for review and comment in advance of any submission, and delay publication, if requested, to allow the Sponsor to preserve its proprietary rights.